CLINICAL TRIAL: NCT06925893
Title: Lutein by Scleral Iontophoresis in Patients With Stage 3 Age-Related Macular Degeneration
Brief Title: Lutein by Scleral Iontophoresis in AMD
Status: Recruiting | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Ciro Costagliola, director, Federico II University
Other Study IDs: 05809854 Federico II; Federico II university (Registry Identifier: Federico II university)
Record Dates: First submitted 2025-03-20; First posted 2025-04-13 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Stage 3 AMD
Keywords: Lutein; AMD; Ionto retina

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of the clinical investigation is to evaluate the performance, safety and degree of tolerability resulting from the use of the iontophoresis medical device in adult subjects diagnosed with AMD stage 3 (AREDS classification) in one or both eyes.

DETAILED DESCRIPTION:
Lutein is a dietary carotenoid which, together with its isomer zeaxanthin, is the main component of the macular pigment of the retina.

Clinical studies have shown that prolonged oral lutein supplementation is safe and is associated with a reduction in the risk of progression from early to advanced stages of Age-Related Macular Degeneration (AMD). However, patient compliance, due to daily oral intake of lutein tablets for a prolonged period of life, is still limited. Additionally, an obstacle to oral supplementation is the variable absorption of lutein through the digestive route.

An iontophoresis method for conveying substances into the eye has been known for some time and already used in the treatment of keratoconus. In this case the substance conveyed is Riboflavin.

A medical device is now available with the following intended use: to combat all oxidative pathologies of the retina and macula, and in particular in the prevention of AMD and in the management of the patient during the evolution of the pathology.

The device consists of an iontophoresis system with scleral applicator and an ophthalmic liquid lutein solution, both of which have already obtained the CE mark. The system therefore includes a generator called K-IONO (CE in class IIa) and a kit called IONTORETINA, which includes a sterile 2 ml vial of lutein (CE in class IIb), the forward and return electrode . which consists of a scleral iontophoresis applicator and an ophthalmic liquid solution of lutein. The topical application of lutein has the advantage of improving the patient's compliance with lutein supplementary therapy compared to oral intake of the carotenoid; Furthermore, in situ application would allow high (therapeutic) concentrations of lutein to be reached in the macular area in a very short period of time (hours) compared to oral intake (months). Publicly available clinical data on scleral iontophoresis or lutein supplementation have not demonstrated any safety-related adverse events and at the same time have demonstrated a reduction in the cumulative risk of progression of AMD from intermediate to advanced stages of the disease.

The objective of the clinical investigation is to evaluate the performance, safety and degree of tolerability resulting from the use of the iontophoresis medical device in adult subjects diagnosed with AMD stage 3 (AREDS classification) in one or both eyes.

ELIGIBILITY:
Inclusion Criteria:

Subjects (male or female) aged ≥ 55 years; Subject able to provide Informed Consent, in compliance with good clinical practice and current legislation

Subject with age-related macular degeneration (AMD) category 3 in one or both eyes classified according to the criteria reported by "Age-Related Eye Disease Study (AREDS)" based on clinical manifestations:

Subject in good general health; Manifest spherical equivalent refraction between +4.0 diopters (D) and - 4.0 D; Best corrected visual acuity (BCVA) for glasses ≤ 0.1 LogMAR; Intraocular pressure (IOP) ≤ 20 mmHg; Subjects able to cooperate with the Investigator; Subjects able to meet the requirements of the entire clinical investigation; Subject who qualifies for treatment with Iontoretina according to the approved indication;

Exclusion Criteria:

Ocular surgery or other type of invasive intervention within the previous 3 months (of any type, including laser surgery and intravitreal injections) performed on the study eye; Lesions, scars, or abrasions of the ocular components present in the eye under study; Dense opacities of the ocular components of the study eye; Implantation of intraocular lenses (IOLs) in the study eye; Congenital malformations in the study eye; Medical history of ocular hypertension and glaucoma, macular pucker, optic neuropathy, diabetic retinopathy, dry eye syndrome, etc. (limited to the study eye);

Lutein or zeaxanthin supplementation or any supplementation or with the intention of impacting eye health within the last 4 weeks prior to the screening visit; Known or potential allergy or hypersensitivity and/or history of allergic reactions to any of the components of the medical device or other chemically closely related substances; Subject suffering from type I diabetes, or with a previous case of stroke; Subject suffering from uncontrolled hypertension and heart disease that, in the opinion of the Investigator, does not allow participation in the study or could compromise the results; Subject smoker (more than 20 cigarettes per day); Significant alcohol consumption: more than 2 drinks per day;

Women of childbearing potential will be excluded from participation in the study if they meet any of the following conditions:

pregnant; intend to become pregnant during the study treatment period; Concomitant hormone replacement therapy for menopause. Participation in another clinical study within the previous 90 days; Subject unable to follow clinical investigation procedures and follow-up visits;

Ages: 55 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects (male or female) aged ≥ 55 years;
  Subject with age-related macular degeneration (AMD) category 3 in one or both eyes classified according to the criteria reported by "Age-Related Eye Disease Study (AREDS)" based on clinical manifestations:
  Subject in good general health; Manifest spherical equivalent refraction between +4.0 diopters (D) and - 4.0 D; Best corrected visual acuity (BCVA) for glasses ≤ 0.1 LogMAR; Intraocular pressure (IOP) ≤ 20 mmHg;
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
BCVA changes [Time Frame: 12 months] Changes in best distance-corrected visual acuity (BCVA) at the End of Study Visit compared to baseline. | 6 months

SECONDARY OUTCOMES:
BCVA changes [Time Frame: 3, 6 and 12 monhs] Changes in best distance-corrected visual acuity (BCVA) at scheduled controls (Visit 3, Visit 4, Visit 5, and Visit 6) compared to baseline | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Federico II University, Naples, Italy

IPD SHARING:
Plan to Share IPD: No